CLINICAL TRIAL: NCT04693143
Title: Parenteral Nutrition for Critically Ill Children
Brief Title: Timing of Initiation of Parenteral Nutrition for Critically Ill Children
Acronym: TPN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Nagwan Yossery Saleh, Assistant professor of Pediatrics, Menoufia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 192119PED14.
Record Dates: First submitted 2020-12-24; First posted 2021-01-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Critical Illness
Keywords: Critically; Pediatric; Parenteral; Nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: A randomized controlled open-label clinical trial
Masking Description: A). Primary outcome for assessment of participants who need mechanical ventilation(MV) and MV duration.
  B). Secondary outcomes will include assessment of participants accordingly, Pediatric Intensive Care Unit (PICU) stay , days of need for vasoacitive drugs infusion , incidence of new infections ,and PICU mortality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parenteral Nutrition for Critically Ill Children (Other): Total Parenteral Nutrition for critically ill children
  Interventions: Other: A randomized controlled open-label clinical trial.

INTERVENTIONS:
Other: A randomized controlled open-label clinical trial. — This was a single-center; open-label randomized controlled trial performed at a Pediatric Intensive Care Unit (PICU) in tertiary care hospital

SUMMARY:
Parenteral Nutrition (PN) is prescribed to children with a non functioning gut. Timing of initiation of PN for critically ill children is a hotly issue. Therefore investigators aim to determine the optimal timing of initiation of PN among these children.This is a randomized clinical trial will be conducted at a Pediatric Intensive Care Unit(PICU) in tertiary care hospital. 140 participants will be randomized to receive either early or late PN. The 1st group gives PN on the 1st day of PICU admissions while the 2nd group gives late PN on the 7th day. Under-nutrition children, early PN will start on the 1st day while late PN begins on 4th day of admission. The outcomes are assessment of mechanical ventilation duration, PICU length stay, and mortality.

DETAILED DESCRIPTION:
Participants and Methods:

This is a single-center; open-label randomized controlled trial will be performed at a Pediatric Intensive Care Unit (PICU) in tertiary care hospital . On admission, patients will be evaluated through history, clinical examination, and investigation.Basic investigations will include complete blood count, serum electrolytes, blood gas analysis, serum creatinine and liver function tests. The severity of the clinical condition upon admission will be determined by calculation of pediatric Sequential Organ Failure Assessment (pSOFA) score and Pediatric Risk of Mortality (PRISM) at the end of the first 24 hours. Patients will be randomized to receive either early or late parenteral nutrition. Early parenteral nutrition will be given in the 1st 24 hours of admission while late parenteral nutrition will be initiated on 7th day of admission. Randomization will be performed by using computer generated random numbers.The patients and the treating physicians will be not blinded to the type of parenteral fluids given. For children with moderate/severe under-nutrition, early parenteral nutrition will start on the 1st day while late parenteral nutrition will on 4th day of admission. This difference in timing of feeding is based on the fact that malnourished children have limited energy reserves and insufficient nutrition for 6 days might be too long a period compared with the case of well-nourished children. Parenteral nutrition consists of glucose, protein, electrolytes (sodium, potassium, calcium, magnesium, and phosphorus), trace elements, water soluble vitamins, and amino acid solutions.Lipid emulsions will be given . The nutritional status of patients will be carefully assessed. The admission weight and length/height will be recorded and a patient will be deemed to have under-nutrition if weight for length z-score is ≤ -2 SD. For children > 36 months, weight/age z-score ≤ -2 SD is used , instead, to define under-nutrition because measuring the height is difficult for critically ill children.

ELIGIBILITY:
Patients' eligibility inclusion criteria:

• Critically ill children admitted to PICU for various reasons and unable to receive their full caloric requirements through the enteral route will be eligible for this study.

Exclusion criteria:

* Included expected short PICU stay < 3 days e.g. Diabetic ketoacidosis;
* Age under 1 month or over 16 years.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Association of timing of Parental nutrition with Need for Mechanical ventilation and its duration. | 3 months
  Need for Mechanical ventilation and duration in days.

SECONDARY OUTCOMES:
Association of timing of Parental nutrition with mortality ,Vasoactive infusion days, and Incidence of new infections. . | 3 months
  Secondary outcomes included: 1).PICU stay in days, 2).Duration of Vasoactive infusion in days; 3). Incidence of new infections; and 4). PICU mortality.
  of new infections; and PICU mortality.

IPD SHARING:
Plan to Share IPD: No
open-label randomized controlled trial performed at a Pediatric Intensive Care Unit (PICU) in tertiary care hospital